CLINICAL TRIAL: NCT05904847
Title: The Effect of Education Given to Diabetes Patients According to the Planned Behavior Theory on Patient Empowerment and Self-Efficacy: A Single-Blind Randomized Controlled Trial
Brief Title: The Effect of Theory-Based Education on Patient Empowerment and Self-Efficacy in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 13353
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Diabete Type 2
Keywords: Diabetes; Theory Of Planned Behavior; Patient Empowerment; Self-Efficacy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Patient Participation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Application of The Theory of Planned Behaviour for Diabetes
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Application of The Theory of Planned Behaviour for Diabetes — In the study, diabetes education consisting of a total of 4 sessions structured according to the Planned Behavior Theory will be applied to the intervention group, and a standard diabetes education consisting of a single session containing information about diabetes on the website of the Ministry of Health will be applied to the control group. The training will be given face-to-face in groups of 10-15 people. After the training, the participants will be monitored for 3 months. To increase patient empowerment and self-efficacy, the intervention group will be followed up by phone calls every 15 days to increase motivation and answer questions.
  Arms: Intervention

SUMMARY:
It is essential to manage the disease to prevent and reduce complications and mortality in patients with diabetes. Adequate information and options should be provided to patients by healthcare providers so that patients can make informed choices. Patient education is a patient empowerment process designed to enable patients to be responsible for their health. With this study, it is considered essential to educate diabetic patients according to the theory of planned behavior and to develop self-efficacy by contributing to patient empowerment in this way.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* 40 years and older
* Diagnosed with type 2 DM at least 1 year ago
* Treated at the hospital where the study will be conducted
* Using antidiabetic agents
* No communication problem
* Contactable by phone

Exclusion Criteria:

* Those who do not meet the inclusion criteria for the study
* Participants who did not give consent at any stage of the study and left

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2023-04-16 (Actual); Primary Completion 2023-06-17 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
Patient Empowerment Scale | 2 weeks
  The scale consists of 37 items in total. Scale is graded in a 5-point Likert type, and in total, the lowest 37 and the highest 185 points are taken. There is an opposite item in the scale. This applied to individuals over the age of 18 who receive long-term care services.
Diabetes Management Self-Efficacy Scale for Patients with Type 2 Diabetes | 2 weeks
  The scale consists of 20 items in total. The scale is scored as a Likert type (1=Never, 2=Rarely, 3=Sometimes, 4=Often, 5=Always), and the lowest score from the scale is 20 and the highest score is 100.

SECONDARY OUTCOMES:
Blood Glucose Level | 3 months
  A condition in which the blood glucose level is above normal. Hyperglycemia is mentioned when fasting blood glucose exceeds 100 mg/dl and postprandial blood glucose exceeds 140 mg/dl.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University, Sakarya, Serdivan, Turkey (Türkiye)

REFERENCES:
- [Derived] Goger S, Sener S, Ci Ngi L D. The effect of training to diabetes patients according to planned behavior theory on self-efficacy and patient empowerment: A randomized study. Prim Care Diabetes. 2024 Oct;18(5):486-492. doi: 10.1016/j.pcd.2024.08.002. Epub 2024 Aug 24. PMID 39183095